CLINICAL TRIAL: NCT07298616
Title: The Efficacy and Safety of the Huaxi Tunnel Technique for Exposure and Dissection of the Recurrent Laryngeal Nerve in Thyroid Surgery：A Prospective, Single-Blind, Randomized Controlled Clinical Study
Brief Title: Huaxi Tunnel Technique For Recurrent Laryngeal Nerve Exposure And Dissection In Thyroid Surgery
Acronym: Huaxi Tunnel
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: West China Hospital (Other)
Collaborators: West China Tianfu Hospital, Sichuan University (Unknown); Shang Jin Hospital of West China Hospital,Sichuan University (Unknown); Sun Yat-sen University Cancer Center (SUSUCC) (Unknown); Sichuan Provincial People's Hospital (Other); Sanya People's Hospital (Unknown)
Responsible Party: Principal Investigator, Yu Feng, West China Hospital, Sichuan University, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024（2498）
Record Dates: First submitted 2025-11-22; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Patients Undergoing Open Thyroid Surgery
Keywords: thyroid surgery; recurrent laryngeal nerve; Huaxi tunnel technique; epinephrine
MeSH Terms: interventions — Epinephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Huaxi Tunnel Technique Group (Experimental): Experimental group (Huaxi tunnel technique group):
  A 5-ml syringe was loaded with adrenaline solution diluted in normal saline (1 mg adrenaline in 250 ml saline, concentration 4 µg/ml) and fitted with a 2-3 cm soft extension tube as the injection tip. After the recurrent laryngeal nerve (RLN) was identified by the cross-hatch method at the posteroinferior capsule below the lower pole of the thyroid gland, the solution was rapidly injected along the RLN's course toward its laryngeal entry point. The hydraulic pressure created by this rapid injection separated the fibrous connective tissue surrounding the nerve, forming a tissue tunnel from the initial identification site to the laryngeal entry point. Subsequent nerve dissection was then performed within this tunnel.
  Interventions: Procedure: Huaxi Tunnel Technique
- Control group (No Intervention): Control group (conventional group): the group in which the recurrent laryngeal nerve was exposed and the thyroid gland was resected by standard thyroid surgical techniques.

INTERVENTIONS:
Procedure: Huaxi Tunnel Technique — A 5-ml syringe was loaded with adrenaline solution diluted in normal saline (1 mg adrenaline in 250 ml saline, concentration 4 µg/ml) and fitted with a 2-3 cm soft extension tube as the injection tip. After the recurrent laryngeal nerve (RLN) was identified by the cross-hatch method at the posteroinferior capsule below the lower pole of the thyroid gland, the solution was rapidly injected along the RLN's course toward its laryngeal entry point. The hydraulic pressure created by this rapid injection separated the fibrous connective tissue surrounding the nerve, forming a tissue tunnel from the initial identification site to the laryngeal entry point. Subsequent nerve dissection was then performed within this tunnel.
  Other Names: adrenaline
  Arms: Huaxi Tunnel Technique Group

SUMMARY:
Protection of the recurrent laryngeal nerve (RLN) is a key focus and difficulty in thyroid surgery. Unilateral RLN injury can lead to ipsilateral vocal cord paralysis, resulting in hoarseness in patients postoperatively. Bilateral RLN injury, however, may cause bilateral vocal cord paralysis, leading to dyspnea and even asphyxiation; in severe cases, tracheotomy and permanent tracheal cannulation are required. Consequently, RLN injury significantly impacts patients' postoperative quality of life and career development. Guidelines and consensuses both domestically and internationally recommend that during the management of the posterior thyroid capsule, active detection, exposure, and dissection of the RLN, combined with meticulous capsular dissection along the RLN, should be performed to effectively reduce the incidence of RLN injury. While active anatomical identification of the RLN can clarify the nerve branches and their relationship with surrounding tissues, facilitating surgical procedures such as ligation and hemostasis, the traditional method of dissecting with instruments like hemostats or right-angle forceps (either blunt or sharp dissection along the nerve surface) increases the risk of nerve injury due to traction, clamping, or thermal damage. This is particularly challenging for less experienced surgeons, who face great difficulties in using energy devices near the RLN without causing injury-a major concern in the field of thyroid surgery.

Diluted epinephrine solution exhibits excellent hemostatic effects in local surgery, improves surgical field clarity, and shortens operation time. Its safety has been clinically verified, and it is commonly used in plastic and cosmetic surgery, joint surgery, and the cavity creation process of endoscopic thyroid surgery. Based on this, this study innovatively proposes the "Huaxi Tunnel Technique": on the basis of meticulous posterior capsular dissection in traditional thyroid surgery, the RLN detection point on the posterior capsule below the lower pole of the thyroid is located using the "cross method" and exposed. A syringe containing diluted epinephrine solution is then used, with its front hose inserted along the RLN towards the laryngeal entry direction. Rapid injection is performed, and the pressure generated by this injection separates the fibrous connective tissue on the RLN surface, forming a "tunnel" from the RLN detection point to the laryngeal entry site-thus achieving exposure and dissection of the RLN.

This technique offers multiple advantages: epinephrine reduces local bleeding, enhancing surgical safety and the convenience of meticulous capsular dissection; tunnel formation causes edema and discoloration of the fibrous connective tissue in the posterior thyroid capsule (while the parathyroid glands remain uncolored), facilitating the rapid identification and protection of the parathyroid glands. Preliminary preclinical experiments have confirmed that the technique reduces the difficulty of RLN exposure and dissection, decreases intraoperative bleeding and complication rates, and improves the safety of thyroid surgery. To further evaluate the efficacy, safety, and operability of this tunnel technique for RLN exposure and dissection, a prospective single-blind randomized controlled trial comparing it with traditional thyroid surgery methods is hereby conducted.

DETAILED DESCRIPTION:
This study is a multicenter, single-blind, randomized controlled trial. Eligible patients will be randomly assigned in a 1:1 ratio to either the experimental group (Tunnel Method group) or the control group (Traditional Method group).

ELIGIBILITY:
Inclusion Criteria:

Aged 18-75 years, regardless of gender Patients hospitalized for open thyroid surgery (undergoing at least unilateral lobe and isthmus resection) and undergoing the procedure for the first time Preoperative color Doppler or contrast-enhanced ultrasound assessment indicates no significant invasion of the recurrent laryngeal nerve by the lesion Participants voluntarily agree to join the trial and provide signed informed consent.

Exclusion Criteria:

History of thyroid nodule ablation therapy Patients scheduled for lateral neck dissection History of hypertension, atrial fibrillation, or severe arrhythmia Uncontrolled subacute thyroiditis or hyperthyroidism Severe comorbidities affecting major organs (cardiac, pulmonary, hepatic, or renal) Presence of cancer-related cachexia syndrome History of psychiatric disorders or cognitive impairment Pregnant or lactating women Participation in other clinical trials within 90 days Other conditions deemed by investigators as unsuitable for trial participation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Recurrent laryngeal nerve injury signal amplitude | Intraoperative
  Differences in nerve signal amplitude before and after RLN dissection at 1 mA and 3 mA.
Assessment of bleeding during RLN dissection | Intraoperative
  After the nerve is identified, a dry gauze is placed; the difference in gauze weight before and after nerve dissection is used to quantify blood loss.
Duration of RLN dissection | Intraoperative
  The time point immediately before and immediately after nerve dissection are recorded, and the interval is calculated as the time required for RLN dissection.
Assessment of parathyroid gland identification and preservation | Preoperative, Intraoperative, 1 day postoperative, 1 month postoperative
  The evaluation is carried out in four domains: (1)Vascularity of the preserved parathyroid glands;(2) Surgeon's subjective rating of parathyroid recognizability during operation (poor / fair / good);(3) Intra-operative autotransplantation of parathyroid tissue (number of fragments transplanted);(4)Change in serum PTH and calcium levels from pre-operative to post-operative measurements
VHI-10 | The day before surgery, 1 day postoperative
  A voice disorder index scale consisting of 10 items, including 5 functional items, 3 physical items, and 2 emotional items. Each item is scored from 0 to 4, with different scores representing the frequency of occurrence: "never" = 0; "rarely" = 1; "sometimes" = 2; "often" = 3; and "always" = 4. A higher score indicates a greater impact of voice disorders on that aspect and a more severe self-assessment of voice impairment. The critical value for VHI is 8 points, and individuals with a VHI score ≥ 8 are considered to have voice dysfunction. Patients need to complete the VHI-10 questionnaire before surgery and on the first day after surgery.
V-RQOL questionnaire | The day before surgery, 1 day postoperative
  Voice-Related Quality of Life-10 (V-RQOL-10): Comprising 10 items, it includes two dimensions: social-emotional and physical-functional. The content of the items describes the subjective experiences of patients with voice disorders. Severity is rated on a scale of 1 to 5, where 1 represents "not at all," 2 represents "a little," 3 represents "a moderate amount," 4 represents "a lot," and 5 represents "extremely." This questionnaire uses "reverse scoring" and must ultimately be converted to a range of 0 to 100 points. A higher overall score indicates better voice quality, while a lower score indicates poorer voice quality.Patients need to complete the V-RQOL questionnaire before surgery and on the first day after surgery.

SECONDARY OUTCOMES:
Total operative time | Intraoperative
  The interval from skin incision to skin closure is recorded to evaluate the impact of the different surgical techniques on overall procedure length.
Postoperative drainage volume | 1 day postoperative, 2 days postoperative, 3 days postoperative, 4 days postoperative
  The total drain output before removal is recorded to assess the impact of the different surgical techniques on overall postoperative drainage.
Blood Pressure | The day before surgery, Intraoperative, 1 day postoperative
  Pre-operative and first post-operative day systolic/diastolic blood pressure are recorded, together with the highest intra-operative BP values, to evaluate side-effects of topical epinephrine use.
  Baseline data including history of hypertension is also registered.
Assessment of local epinephrine-related adverse effects | The day before surgery, Intraoperative, 1 day postoperative
  Pre-operative and first post-operative day heart rate is recorded, together with the highest intra-operative HR values, to evaluate side-effects of topical epinephrine use.
  Baseline data including history of arrhythmia is also registered.
Assessment of local epinephrine-related adverse effects | 1 day postoperative
  Any post-operative symptoms are documented: palpitations, headache, elevated BP, tremor, weakness, dizziness, vomiting, cold extremities, arrhythmia or ventricular fibrillation.

CONTACTS AND LOCATIONS:
Locations (1):
- West China hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] GBD 2019 Diseases and Injuries Collaborators. Global burden of 369 diseases and injuries in 204 countries and territories, 1990-2019: a systematic analysis for the Global Burden of Disease Study 2019. Lancet. 2020 Oct 17;396(10258):1204-1222. doi: 10.1016/S0140-6736(20)30925-9. PMID 33069326
- [Result] Haymart MR. Progress and Challenges in Thyroid Cancer Management. Endocr Pract. 2021 Dec;27(12):1260-1263. doi: 10.1016/j.eprac.2021.09.006. Epub 2021 Sep 22. PMID 34562612